CLINICAL TRIAL: NCT06781008
Title: Emerging Tick-borne Diseases in Children and Adults in Sweden (SWEtick): a Prospective Multicenter Study for Improved Patient Management
Brief Title: SWEtick - a Prospective Multicenter Study of Tick-borne Diseases in Sweden
Status: Recruiting | Type: Observational
Sponsor: Anna J Henningsson (Other Government)
Collaborators: Region Östergötland (Other); Region Kalmar County (Unknown); Region Dalarna (Unknown); FORSS - The Research Council of South-Eastern Sweden (Unknown); ALF Grants, Region Östergötland (Unknown); Linkoeping University (Other Government)
Responsible Party: Sponsor-Investigator, Anna J Henningsson, Senior Consultant, Senior Associate Professor, Region Jönköping County
Organization: Region Jönköping County (Other Government)
Other Study IDs: EPM 2022-05330-01
Record Dates: First submitted 2025-01-08; First posted 2025-01-17 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Tick-Borne Diseases
MeSH Terms: conditions — Tick-Borne Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Whole blood, skin biopsies, cerebrospinal fluid, synovial fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- TBD: Patients with confirmed tick-borne disease
- Non-TBD: Patients investigated for suspected tick-borne disease but diagnosed with another condition (tick-borne disease excluded)
- Control group CNS: Patients obtaining spinal anasthesia in conjunction with knee or hip replacement surgery due to arthrosis
- Control group arthritis: Patients with autoinflammatory joint disease
- Control group healthy: Blood donors

SUMMARY:
The purpose of the SWEtick project is to increase the knowledge of the various clinical presentations of emerging tick-borne diseases (eTBD), to assess their importance for human health, to develop and validate laboratory methods for diagnosis of eTBD, and to develop recommendations for knowledge-driven management of patients with suspected eTBD within the Swedish healthcare system.

ELIGIBILITY:
Inclusion Criteria in TBD and Non-TBD groups:

* Clinical suspicion of tick-borne disease (physician's assessment based on medical history, symptoms, clinical findings and sometimes laboratory results)

Exclusion Criteria:

* Incapacitated to understand the study information and make decisions (adults and adolescents >15 years)

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Medical history: tick exposure, tick bite, splenectomy, immunosuppressive treatment (e.g. anti-CD20 or other biological/immunomodulatory drugs, cortisone corresponding to >10 mg prednisolone/day, chemotherapy, hematologic malignancy, other malignancy, rheumatologic disease)
  2. Symptoms/clinical signs: fever after tick bite, relapsing fever of unknown origin, skin rashes (single/multiple erythema migrans, lymphocytoma, acrodermatitis chronica atrophicans or other), venous thrombosis, repeated thrombophlebitis, meningitis, encephalitis, myelitis, cranial nerve palsy, radiculitis, peripheral nerve involvment, mono-/oligoarthritis, carditis, ocular or otogenic disturbances of uncertain origin where medical history includes recent tick bite.
  3. Biochemical findings in combination with factors under a) and b): leukopenia, thrombocytopenia, anemia, elevated liver enzymes, slightly elevated erythrocyte sedimentation rate and/or C-reactive protein, pleocytosis in CSF or synovial fluid.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
EuroQoL-5 Dimension Questionnaire (EQ-5D) | 6 months
  Difference in EQ-5D Health index between study inclusion and at the 6 month-follow-up
Visual Analogue Scale for Health (VAS) | 6 months
  Difference between the VAS units at study inclusion and at 6 month-follow-up.

CONTACTS AND LOCATIONS:
Locations (6):
- Sweden (6):
  - Department of Paediatrics, Eksjö Hospital, Eksjö, Region Jönköping County
  - Department of Infectious Diseases, County Hospital Ryhov, Jönköping, Region Jönköping County
  - Department of Infectious Diseases, Kalmar County Hospital, Kalmar, Region Kalmar County
  - Department of Infectious Diseases, Linköping University Hospital, Linköping, Region Östergötland
  - Department of Infectious Diseases, Vrinnevi Hospital, Norrköping, Region Östergötland
  - Department of Paediatrics, Vrinnevi Hospital, Norrköping, Region Östergötland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication can be shared after anonymization, upon request

REFERENCES:
- [Background] Henningsson AJ, Asgeirsson H, Hammas B, Karlsson E, Parke A, Hoornstra D, Wilhelmsson P, Hovius JW. Two Cases of Borrelia miyamotoi Meningitis, Sweden, 2018. Emerg Infect Dis. 2019 Oct;25(10):1965-1968. doi: 10.3201/eid2510.190416. PMID 31538916
- [Background] Uhnoo I, Cars O, Christensson D, Nystrom-Rosander C. First documented case of human babesiosis in Sweden. Scand J Infect Dis. 1992;24(4):541-7. doi: 10.3109/00365549209052642. PMID 1411322
- [Background] Eimer J, Fernstrom L, Rohlen L, Grankvist A, Loo K, Nyman E, Henningsson AJ, Haglund M, Hultqvist V, Sjowall J, Wenneras C, Schon T. Spiroplasma ixodetis Infections in Immunocompetent and Immunosuppressed Patients after Tick Exposure, Sweden. Emerg Infect Dis. 2022 Aug;28(8):1681-1685. doi: 10.3201/eid2808.212524. PMID 35876734
- [Background] Bjoersdorff A, Berglund J, Kristiansen BE, Soderstrom C, Eliasson I. [Varying clinical picture and course of human granulocytic ehrlichiosis. Twelve Scandinavian cases of the new tick-borne zoonosis are presented]. Lakartidningen. 1999 Sep 29;96(39):4200-4. Swedish. PMID 10544585
- [Background] Nilsson K, Elfving K, Pahlson C. Rickettsia helvetica in patient with meningitis, Sweden, 2006. Emerg Infect Dis. 2010 Mar;16(3):490-2. doi: 10.3201/eid1603.090184. PMID 20202426
- [Background] Nilsson K, Lindquist O, Pahlson C. Association of Rickettsia helvetica with chronic perimyocarditis in sudden cardiac death. Lancet. 1999 Oct 2;354(9185):1169-73. doi: 10.1016/S0140-6736(99)04093-3. PMID 10513711
- [Background] Wenneras C, Wass L, Bergstrom B, Grankvist A, Lingblom C. Ten years of detecting Neoehrlichia mikurensis infections in Sweden: demographic, clinical and inflammatory parameters. Eur J Clin Microbiol Infect Dis. 2024 Nov;43(11):2083-2092. doi: 10.1007/s10096-024-04909-5. Epub 2024 Aug 13. PMID 39136831
- [Background] Quarsten H, Henningsson A, Krogfelt KA, Strube C, Wenneras C, Mavin S. Tick-borne diseases under the radar in the North Sea Region. Ticks Tick Borne Dis. 2023 Jul;14(4):102185. doi: 10.1016/j.ttbdis.2023.102185. Epub 2023 Apr 26. PMID 37116420
- [Background] Henningsson AJ, Aase A, Bavelaar H, Flottorp S, Forsberg P, Kirkehei I, Lovmar M, Nilsson K, Nyman D, Ornstein K, Sjowall J, Skogman BH, Tjernberg I, Aaberge I. Laboratory Methods for Detection of Infectious Agents and Serological Response in Humans With Tick-Borne Infections: A Systematic Review of Evaluations Based on Clinical Patient Samples. Front Public Health. 2021 Sep 20;9:580102. doi: 10.3389/fpubh.2021.580102. eCollection 2021. PMID 34616701
- See also: General study information and contact details — https://liu.se/forskning/fastingburna-infektioner/swetick